CLINICAL TRIAL: NCT04989127
Title: Comparison The Postoperative Effects Of Local Antibiotic Versus Systemic Antibiotic With The Use Of Platelet Rich Fibrin On The Mandibular Third Molar Surgery
Brief Title: Comparison The Postoperative Effects of Local and Systemic Antibiotics Applied With Platelets Rich Fibrin
Status: Completed | Type: Observational
Sponsor: Ceren Melahat Donmezer (Other)
Responsible Party: Sponsor-Investigator, Ceren Melahat Donmezer, Phd student, Near East University, Turkey
Organization: Near East University, Turkey (Other)
Other Study IDs: YDU/2019/67-774
Record Dates: First submitted 2021-07-01; First posted 2021-08-04 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Impacted Wisdom Tooth
Keywords: platelets rich fibrin; systemic antibiotic; local antibiotic; comparison
MeSH Terms: interventions — Diagnosis; Penicillins; Analgesics; Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- group 1: platelet-rich fibrin placed into the socket of the extracted tooth.+ Augmentin 1 gr tablet prescribed 3 times a day
  Interventions: Diagnostic Test: Diagnosis; Procedure: traditional osteotomies; Biological: Platelet Rich Fibrin; Drug: Antibiotics, Penicillin; Drug: Analgesic
- group 2: platelet-rich fibrin + 0.5 ml amoklavin I.V. 1.2 gr placed into the socket of the extracted tooth.
  Interventions: Diagnostic Test: Diagnosis; Procedure: traditional osteotomies; Biological: Platelet Rich Fibrin; Drug: Antibiotics, Penicillin; Drug: Analgesic
- group 3: platelet-rich fibrin placed into the socket of extracted tooth + Clin 150 mg capsule prescribed 4 times a day
  Interventions: Diagnostic Test: Diagnosis; Procedure: traditional osteotomies; Biological: Platelet Rich Fibrin; Drug: Analgesic; Drug: Antibiotic
- group 4: platelet-rich fibrin + 0.5 ml Clin 600 mg/4 ml IM/IV, 0.5 ml placed into the socket of the extracted tooth.
  Interventions: Diagnostic Test: Diagnosis; Procedure: traditional osteotomies; Biological: Platelet Rich Fibrin; Drug: Analgesic; Drug: Antibiotic
- control group: platelet-rich fibrin placed into the socket of extracted tooth and no antibiotic is prescribed.
  Interventions: Diagnostic Test: Diagnosis; Procedure: traditional osteotomies; Biological: Platelet Rich Fibrin; Drug: Analgesic

INTERVENTIONS:
Diagnostic Test: Diagnosis — All of the patients withstand a radiological examination, including panoramic radiography, and all were handled by the same surgeon and assistant.
Procedure: traditional osteotomies — In all groups the flap incision was triangular in shape which avoids muscle involvement (Archer flap).
Biological: Platelet Rich Fibrin — Platelet rich fibrin (PRF), is an example and popular procedure for accelerate healing of soft and hard tissue because of the presence of various growth factors.a blood sample was taken without anticoagulant in 10 mL glass-coated plastic tubes that were immediately centrifuged (Elektro-mag M415P) at 3,000 rpm for 10 min (approximately 400 g) (13). The platelet-poor plasma that accumulated at the top of the tubes was discarded.PRF was dissected approximately 2 mm below its contact point with the red corpuscles situated beneath, to include any remaining platelets that may have localized below the junction between the PRF and red corpuscles.
Drug: Antibiotics, Penicillin — Antibiotics are prescribed for the patients.
  Groups: group 1; group 2
Drug: Analgesic — Analgesics are prescribed for the patients.
Drug: Antibiotic — Patients with penicillin allergy
  Groups: group 3; group 4

SUMMARY:
The aim of this study was investigate the comparison of postoperative effects of local antibiotics mixed with platelet-rich fibrin and postoperative systemic antibiotic applications prescribed for mandibular impacted third molar tooth extraction. The study included a total of 75 patients with impacted mandibular third molar. Patients were evaluated in 5 randomly separated groups. For the first and third group, Platelets Rich Fibrin+ systemic Antibiotics were applied into the tooth socket and for the second and fourth group, Platelets Rich Fibrin + local antibiotics were applied, respectively. There was a control group which only Platelets Rich Fibrin was applied into the socket. The outcome variables were pain, swelling, the number of analgesics taken, and trismus. These variables were also assessed based on first, second, third, and seventh days following the operation.

ELIGIBILITY:
Inclusion Criteria:

* The patient had no systemic diseases, no taken opioids for a long period, no current infections or acute pericoronitis, no smoke or drink alcohol, no pregnancy, the absence of allergy to penicillin and presence of penicillin allergy.

Exclusion Criteria:

* pericoronitis, no inflammation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community aged between 18-40 without any important systemic disease.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2019-03-17 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-21 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) | day 1
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
visual analogue scale (VAS) | day 2
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
visual analogue scale (VAS) | day 3
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
visual analogue scale (VAS) | day 7
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
visual analogue scale (VAS) | day 15
  It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.
Trismus | day 1
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | day 2
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | day 3
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | day 7
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
Trismus | day 15
  Trismus by measuring the distance between the mesial incisal corners of the upper and lower right incisors during maximum mouth opening.
swelling | day 1
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
swelling | day 2
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
swelling | day 3
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
swelling | day 7
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.
swelling | day 15
  measured using a flexible plastic measuring tape as described by Gabka and Matsumura by measuring the distance from the corner of the mouth to the attachment of the earlobe following the bulge of the cheek and the distance from the outer canthus of the eye to the angle of the mandible.

OTHER OUTCOMES:
the number of analgesic tablets | day 1,2,3,7 and 15
  Check the patients analgesic number of days 1,2,3,7 and 15.
the number of analgesic tablets | day 2
  Check the patients analgesic number of days 1,2,3,7 and 15.
the number of analgesic tablets | day 3
  Check the patients analgesic number of days 1,2,3,7 and 15.
the number of analgesic tablets | day 7
  Check the patients analgesic number of days 1,2,3,7 and 15.
the number of analgesic tablets | day 15
  Check the patients analgesic number of days 1,2,3,7 and 15.

CONTACTS AND LOCATIONS:
Overall Officials: Ceren Melahat Dönmezer, Principal Investigator — Near East University
Locations (1):
- Near east University, Nicosia, Lefkosa, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polak D, Clemer-Shamai N, Shapira L. Incorporating antibiotics into platelet-rich fibrin: A novel antibiotics slow-release biological device. J Clin Periodontol. 2019 Feb;46(2):241-247. doi: 10.1111/jcpe.13063. PMID 30629300
- [Background] Osunde OD, Adebola RA, Omeje UK. Management of inflammatory complications in third molar surgery: a review of the literature. Afr Health Sci. 2011 Sep;11(3):530-7. PMID 22275950
- [Background] Kreutzer K, Storck K, Weitz J. Current evidence regarding prophylactic antibiotics in head and neck and maxillofacial surgery. Biomed Res Int. 2014;2014:879437. doi: 10.1155/2014/879437. Epub 2014 Jul 8. PMID 25110703
- [Background] Uyanik LO, Bilginaylar K, Etikan I. Effects of platelet-rich fibrin and piezosurgery on impacted mandibular third molar surgery outcomes. Head Face Med. 2015 Jul 26;11:25. doi: 10.1186/s13005-015-0081-x. PMID 26209242